CLINICAL TRIAL: NCT03267732
Title: A Phase 1 Study to Evaluate the Pharmacokinetics of Single and Multiple Doses of AM0010 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics in Participants After Dosing With Pegilodecakin (LY3500518)
Acronym: Willow 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: ARMO BioSciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17297; J1L-AM-JZGE (Other: Eli Lilly and Company); AM0010-801 (Other: ARMO BioSciences)
Record Dates: First submitted 2017-08-24; First posted 2017-08-30 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Healthy Adult Subjects
MeSH Terms: interventions — pegilodecakin; AM0010

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1 (Active Comparator): Pegilodecakin (5 μg/kg) dosed on Day 1, and Days 4-9 SQ
  Interventions: Biological: Pegilodecakin
- 2 (Active Comparator): Pegilodecakin (10 μg/kg) dosed on Day 1, and Days 4-9 SQ
  Interventions: Biological: Pegilodecakin

INTERVENTIONS:
Biological: Pegilodecakin — Pegilodecakin Alone
  Other Names: LY3500518; AM0010

SUMMARY:
To evaluate the pharmacokinetics of single and multiple doses of pegilodecakin in healthy participants.

DETAILED DESCRIPTION:
This is an open-label, single-center, phase 1 study designed to evaluate the pharmacokinetics in healthy adult participants after single and multiple subcutaneous injections of pegilodecakin.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 55 years of age, inclusive
2. Must have a body mass index (BMI) between 19 and 32 (kg/m2) at study Screening
3. Must be HIV negative by HIV 1/0/2 testing
4. Must be Hepatitis B (HBV) surface antigen negative
5. Must be Hepatitis C (HCV) antibody negative
6. Females must have a negative serum pregnancy test
7. Must refrain from blood donation from 30 days prior to Day 0 through completion of the study and continuing for at least 30 days from date of last dose of study drug

Exclusion Criteria:

1. Pregnant or lactating subjects
2. Have previously participated in an investigational trial involving administration of any investigational compound within 30 days prior to the study dosing
3. Have poor venous access and are unable to donate blood
4. Have been vaccinated within 90 days of study dosing
5. Current alcohol or substance abuse judged by the Investigator to interfere with subject compliance
6. Have history of significant drug sensitivity or drug allergy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, Cmax | 43 days
  maximal plasma concentration (Cmax)
Pharmacokinetic parameters, Tmax | 43 days
  maximal concentration (Tmax)
Pharmacokinetic parameters, AUC | 43 days
  area under the plasma concentration curve (AUC)
Pharmacokinetic parameters, CL/F | 43 days
  clearance (CL/F).

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 43 days
  Evaluate the safety of single/multiple SQ doses of Pegilodecakin - Incidence of adverse events, injection site reactions, clinically relevant changes in laboratory values, EKGs, and vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- PPD Development, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No